CLINICAL TRIAL: NCT05605600
Title: A Qualitative Research Study Using Patient Focus Groups to Translate International Consensus Definition of Low Anterior Resection Syndrome (LARS) Into a Bowel Dysfunction Severity Scoring Tool.
Brief Title: Translation of the International Consensus Definition of LARS Into a Bowl Dysfunction Severity Scoring Tool (New LARS Score)
Status: Completed | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: University of Auckland, New Zealand (Other); University of Aarhus (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 8395; 313617 (Other: IRAS); 22/PR/0889 (Other: Wales REC4)
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2022-07

CONDITIONS: Low Anterior Resection Syndrome
Keywords: Qualitative Research; Patient-Reported Outcome Measures; Colorectal Cancer; Bowel Dysfunction
MeSH Terms: conditions — Low Anterior Resection Syndrome; Colorectal Neoplasms; Intestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Low Anterior Resection Syndrome: Patients with lived-experience of anterior resection surgery, who may or may not have subsequently developed bowel dysfunction symptoms, will be invited to take part in a focus group. They will discuss a new questionnaire and the phrasing of the questions, ensuring clarity and reducing the potential variability in interpretation of each question.

SUMMARY:
The purpose of this study is to develop a new severity scoring tool for Low Anterior Resection Syndrome (LARS) drawing on the international consensus criteria for LARS as well as opinions of patients with lived-experience of LARS.

DETAILED DESCRIPTION:
Six out of ten patients have significant bowel problems in the first 12 months after surgery to remove their rectum (last bit of bowel), with as many as 4 out of 10 having longer term issues. This is an operation which is most commonly performed to treat bowel cancer. Bowel problems can include having to rush to the toilet, having accidents or leakage into the underwear or difficulty fully emptying the bowels. This condition is called Low Anterior Resection Syndrome, or 'LARS' for short. The definition of Low Anterior Resection Syndrome was developed in 2020 with patient involvement throughout the process so it accurately captures the real-world experience of LARS. This definition is to be used to create a new scoring system to measure the severity of LARS.

The aim of this study is to transform this new definition into a scoring tool which can be used to assess the severity of Low Anterior Resection Syndrome and investigate how well various treatments work for LARS. It is vital to have patients involved throughout this work to ensure that the new score gives an accurate picture of the severity of these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Able and willing to provide informed consent
* Undergone an anterior resection for cancer, with current bowel continuity

Exclusion Criteria:

* Currently undergoing adjuvant therapy
* Recurrent or metastatic disease
* Unable to participate to complete study procedures (Due to intellectual or cognitive impairment; Due to insufficient English-language skills (oral and written))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of this study is to develop a new scoring tool for Low Anterior Resection Syndrome through patient focus groups. We will identify and recruit patients with lived-experience of anterior resection surgery, who may or may not have subsequently developed bowel dysfunction symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Development of LARS Severity tool | 6 months
  Qualitative research methods will be used develop the new tool. A patient focus group will be conducted to review the draft questionnaire and refine question and response wordings.

SECONDARY OUTCOMES:
Gain patient opinion on new scoring tool name | 6 months
  Focus groups will be asked to rank proposed tool names from 'least favoured' to 'most favoured'. This will be considered along with clinical opinion to derive final tool name.
Commence initial psychometric evaluation of the New LARS score | 6 months
  Participants will be asked to complete the new LARS score tool, along with existing LARS tool to test proposed question set and administration method as well as comparability to existing tool.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Cornish, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- Julie Cornish, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No